CLINICAL TRIAL: NCT01026350
Title: Safety and Efficacy of Oral Colostrum Derived Anti Influenza Antibodies in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Immuron Limited, Immuron Limited
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4811344-HMO-CTIL
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-11

CONDITIONS: Influenza
Keywords: modulating immune response to flu antigen
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- study group (Experimental)
  Interventions: Dietary Supplement: colostrum enriched with anti flu antibodies

INTERVENTIONS:
Dietary Supplement: colostrum enriched with anti flu antibodies — each volunteer will receive six 1.2 g oral tablets (equivalent to 600 mg of bovine colostrum powder each) once a day for two weeks.

SUMMARY:
Administration of colostrum enriched with anti-Flu antibodies may alter host's response to the flu virus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers ages 18-60
* If participating in sexual activity that could lead to pregnancy, the study volunteer must agree that two reliable methods of contraception will be used simultaneously while receiving the protocol-specified medication and for 1 month after stopping the medication
* Men > 18 years.
* Ability and willingness of subject to provide informed consent
* Screening tests' results within 15% of normal values

Exclusion Criteria:

* Female
* Continuous use of the following medications for more than 3 days within 30 days of study entry:
* Immunosuppressives
* Immune modulators
* Systemic glucocorticoids
* Anti-neoplastic agents
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry.
* Subjects with a clinically significant infectious, immune mediated or malignant disease
* Subjects with anemia (Hb <10.5 gm/dl)
* Subjects with thrombocytopenia (platelets <100K/µl)
* Subjects with lymphopenia (absolute lymphocyte count <0.7)
* Subjects who were previously vaccinated against flu.
* Subject who received any vaccination within the last 6 months

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
alterations in immune response to flu antigen | during and after administration of colostrum enriched with anti flu antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Kim JH, Jung WS, Choi NJ, Kim DO, Shin DH, Kim YJ. Health-promoting effects of bovine colostrum in Type 2 diabetic patients can reduce blood glucose, cholesterol, triglyceride and ketones. J Nutr Biochem. 2009 Apr;20(4):298-303. doi: 10.1016/j.jnutbio.2008.04.002. Epub 2008 Jul 7. PMID 18602824